CLINICAL TRIAL: NCT00730002
Title: Magnetic Resonance Spectroscopy, Perfusion, and Diffusion Tensor Imaging in Neuropsychiatric Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Pia C Maly Sundgren, MD, PhD, Primary Investigator, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00000714
Record Dates: First submitted 2008-08-01; First posted 2008-08-08 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Neuropsychiatric Systemic Lupus Erythematosus
Keywords: Lupus
MeSH Terms: conditions — Lupus Vasculitis, Central Nervous System | interventions — Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1- Healthy Subjects (Active Comparator): Healthy Subjects- receive MRA
  Interventions: Procedure: Magnetic Resonance Angiography (MRA); Procedure: Magnetic resonance imaging
- 2 - patients with SLE, no neuropsych (Active Comparator): Systemic Lupus Erythematosus(SLE) patients without neuropsychiatric symptoms - receive MRA
  Interventions: Procedure: Magnetic resonance imaging; Procedure: MRA
- 3 - patients with SLE with neuropsych (Active Comparator): 20 symptomatic neuropsychiatric systemic lupus erythematosus(NPSLE) patients.
  Interventions: Procedure: MRA; Procedure: diffusion Imaging
- 4- healthy patients from other cohort (Active Comparator): 10 Healthy Controls (HC) from an existing cohort as part of another sponsored study.
  Interventions: Procedure: perfusion imaging.

INTERVENTIONS:
Procedure: Magnetic Resonance Angiography (MRA) — As part of the Magnetic Resonance(MR) scan, you will need to lie still on a padded MR table inside the MR machine for about 15 minutes at a time while MR studies are being performed on you. The total time for the clinical portion of the MR study is approximately 35-40 minutes and there will be an additional 30 minutes for the research related MR studies. The total time you will spend on the MR table for this research will seldom be more than one hour.
  Other Names: Magnetic resonance imaging
  Arms: 1- Healthy Subjects
Procedure: Magnetic resonance imaging — MR spectroscopy
  Other Names: MRA
  Arms: 1- Healthy Subjects; 2 - patients with SLE, no neuropsych
Procedure: MRA — MRA of the brain
  Arms: 2 - patients with SLE, no neuropsych
Procedure: MRA
  Arms: 3 - patients with SLE with neuropsych
Procedure: diffusion Imaging — MRA of the Brain
  Arms: 3 - patients with SLE with neuropsych
Procedure: perfusion imaging. — MRA of the brain
  Arms: 4- healthy patients from other cohort

SUMMARY:
The purpose of this study is to determine if three functional Magnetic Resonance brain imaging techniques: Magnetic Resonance Spectroscopy(MRS),Magnetic Resonance perfusion, and Diffusion Tensor Imaging(DTI) can detect brain alterations distinctive for neuropsychiatric systemic lupus erythematosus (NPSLE)and systemic lupus erythematosus(SLE).

DETAILED DESCRIPTION:
Purpose of the Study:

We plan with this study to obtain pilot data to support a larger grant application which will evaluate whether any of three types of functional Magnetic Resonance Imaging (known as MR Spectroscopy [MRS], MR Perfusion Imaging, and MR Diffusion Tensor Imaging [DTI]) can detect alterations in brain function distinctive for Neuropsychiatric Systemic Lupus Erythematosus (NPSLE), Systemic Lupus Erythematosus (SLE), and compare our findings to those found in an existing cohort of 20 normal healthy controls. Because this study is being done on a 3T(tesla)scanner (3T(tesla) Achieva(Model name), Philips Medical Systems) and our previous group of healthy controls was assessed using a 1.5 T(tesla) scanner (LX EchoSpeed, General Electric(GE) Medical Systems), we propose to re-consent 10 of the previous 20 healthy controls and re-collect imaging data on the 3T(tesla) scanner in order to confirm that our previously-collected data from the group of 20 healthy controls is still valid. This will confirm that the change of field strength and manufacturer does not affect data validity.

Recruiting Update as of March/2009: Enrollment is completed for Study Arms 1 and 2.

This study is only being conducted in Ann Arbor, Michigan. Travel reimbursement does not include hotel accommodations or air fare to and from Ann arbor, Michigan.

ELIGIBILITY:
Inclusion Criteria:

* Have no diagnosis of NPSLE, SLE, or any other condition which, in the investigator's opinion, might cause central nervous system(CNS) changes or interfere with the interpretation of results.
* Be 18 years of age or older.
* Be willing and able to complete all study procedures.
* Meet the criteria for diagnosis of systemic lupus erythematosus(SLE).
* Have recent onset or diagnosis of neurological symptoms that have been active within the last 14 days. The criteria for NPSLE study patients will be neurological symptoms, confirmed by neurologic examination, which, in the opinion of the treating physician, may be due to the patient's diagnosis of SLE, and requires MRI evaluation. Patients will be classified according to the nomenclature recommended by the American College Rheumatology(ACR) on Neuropsychiatric Manifestations in SLE, and further classified as "focal," "nonfocal," or "seizure" (64).
* Be able to complete all study procedures; and be able to sign the informed consent form or have a designated proxy or next-of-kin present to provide consent on behalf of the subject.
* Meet the American College of Rheumatology(ACR) criteria for SLE and be a member of the U of M lupus cohort.
* Report no neurological symptoms at the time of enrollment.

Exclusion criteria:

* Co-morbid medical illnesses capable of causing a worsening of physical functional status independent of the diagnosis (e.g. morbid obesity, autoimmune diseases other than SLE), cardiopulmonary disorders (e.g. angina, congestive heart failure, chronic obstructive pulmonary disease(COPD), chronic asthma), fibromyalgia(FM), uncontrolled endocrine or allergic disorders (e.g. thyroid dysfunction, Type I diabetes), and malignancy within 2 years, excluding successfully treated squamous or basal skin carcinoma.
* Any present psychiatric disorder involving a history of psychosis (e.g. schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder etc.), current suicide risk or attempt within 2 years of the study, or substance abuse within 2 years.
* Subjects who are pregnant.
* Subjects who are left-handed.
* Those SLE patients with acute onset of neurological symptoms with duration longer than 14 days.
* Have acute onset of neurological symptoms related to systemic lupus erythematosus(SLE).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-03; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
This pilot data will be used to strengthen our application for a larger grant to definitively study the sensitivity and specificity of these alterations. | At 6 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Pia Maly Sundgren, MD-PHD, Principal Investigator — University of Michigan; Pia Maly Sundgren, MD, PHD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States